CLINICAL TRIAL: NCT00553150
Title: Phase I/II Evaluation of Everolimus (RAD001), Radiation and Temozolomide (TMZ) Followed by Adjuvant Temozolomide and Everolimus in Newly Diagnosed Glioblastoma
Brief Title: Everolimus, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N057K; NCI-2009-00654 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000573917 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult gliosarcoma; adult giant cell glioblastoma; adult glioblastoma; adult anaplastic astrocytoma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult subependymal giant cell astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Gliosarcoma; Glioblastoma; Astrocytoma | interventions — Everolimus; Temozolomide; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (RAD001), Radiation (RT), Temozolomide (TMZ) (Experimental): Patients receive oral everolimus and oral temozolomide and 3D-conformal radiotherapy or IMRT as in phase I. Patients will undergo a 4-6 week rest period in course 2 and then proceed to adjuvant therapy.
  Adjuvant therapy with everolimus and temozolomide (courses 3-8): Patients receive oral everolimus and oral temozolomide as in phase I.
  Adjuvant therapy with everolimus alone (courses 9 and all subsequent courses): Patients receive oral everolimus as in phase I.
  All patients undergo fludeoxyglucose (FDG)- or fluorothymidine-labeled PET/CT scans at baseline and periodically during treatment.
  Interventions: Drug: everolimus; Drug: temozolomide; Radiation: radiation

INTERVENTIONS:
Drug: everolimus
Drug: temozolomide
Radiation: radiation

SUMMARY:
RATIONALE: Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking some of the blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving everolimus together with temozolomide and radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of everolimus when given together with temozolomide and radiation therapy in treating patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose (MTD) of everolimus in combination with temozolomide and 3D-conformal radiotherapy or intensity-modulated radiotherapy (IMRT) followed by adjuvant temozolomide with or without everolimus in patients with newly diagnosed glioblastoma. (Mayo Clinic Rochester [MCR] AND Mayo Clinic Jacksonville [MCJ] patients only) (Phase I)
* To assess and describe the adverse events of everolimus in combination with temozolomide and 3D-conformal radiotherapy or IMRT followed by adjuvant temozolomide with or without everolimus in patients with newly diagnosed glioblastoma. (MCR and MCJ patients only) (Phase I)
* To assess treatment effectiveness of everolimus in combination with temozolomide and 3D-conformal radiotherapy or IMRT followed by adjuvant temozolomide with or without everolimus, until progression, in patients with newly diagnosed glioblastoma. (all North Central Cancer Treatment Group [NCCTG] patients) (Phase II)
* To characterize the toxicities of everolimus in combination with temozolomide and 3D-conformal radiotherapy or IMRT followed by adjuvant temozolomide with or without everolimus in patients with newly diagnosed glioblastoma. (all NCCTG patients) (Phase II)
* Evaluate whether suppression of fludeoxyglucose F18 (18FDG) uptake in tumor and normal brain can be used to determine a biologically effective dose for efficient penetration of everolimus through the blood-brain barrier. (MCR and MCJ patients only) (Phase I)
* Correlate everolimus levels with 18FDG uptake suppression in tumor and normal brain. (MCR and MCJ patients only) (Phase I)
* Assess the relationship between efficacy endpoints (i.e., survival, progression-free survival, and response) and changes in 3'-deoxy-3'-[18F]fluorothymidine (18F-FLT) uptake for patients treated at MCR. (all NCCTG patients) (Phase II)
* Assess the relationship between efficacy endpoints (i.e., survival, progression-free survival, and response), and phospho-Akt, PTEN status, and MGMT expression and promoter methylation status. (all NCCTG patients) (Phase II)
* Assess the relationship between efficacy endpoints (i.e., survival, progression-free survival, and response) and baseline gene expression signatures from paraffin embedded pre-treatment tumor samples. (all NCCTG patients) (Phase II)
* Correlate gene expression between paraffin and frozen samples. (all NCCTG patients) (Phase II)
* Evaluate potential mechanisms of therapy resistance in recurrent tumor samples obtained at the time of surgery for recurrent disease. (Phase I and II)

OUTLINE: This is a multicenter, phase I dose-escalation study of everolimus followed by a phase II study.

* Phase I (Mayo Clinic Rochester [MCR] AND Mayo Clinic Jacksonville [MCJ] ONLY):

  * Concurrent therapy (courses 1 and 2): Patients receive oral everolimus once weekly in weeks 1-7 or 1-8 and oral temozolomide once daily in weeks 2-7 or 3-8. Patients also undergo radiotherapy 5 days a week in either weeks 2-7 or 3-8. Four to six weeks later, patients proceed to adjuvant therapy. This rest period is defined as course 2.
  * Adjuvant therapy with everolimus and temozolomide (courses 3-8): Patients receive oral everolimus on days 1, 8, 15, and 22 and oral temozolomide on days 1-5. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Adjuvant therapy with everolimus alone (courses 9 and all subsequent courses): Patients receive oral everolimus on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression our unacceptable toxicity.
* Phase II (Open to MCR center ONLY) (All North Central Cancer Treatment Group [NCCTG] centers closed to accrual as of 02/17/11):

  * Concurrent therapy (courses 1 and 2): Patients receive oral everolimus and oral temozolomide and 3D-conformal radiotherapy or IMRT as in phase I. Patients will undergo a 4-6 week rest period in course 2 and then proceed to adjuvant therapy.
  * Adjuvant therapy with everolimus and temozolomide (courses 3-8): Patients receive oral everolimus and oral temozolomide as in phase I.
  * Adjuvant therapy with everolimus alone (courses 9 and all subsequent courses): Patients receive oral everolimus as in phase I.

All patients undergo fludeoxyglucose (FDG)- or fluorothymidine-labeled PET/CT scans at baseline and periodically during treatment.

Patients undergo blood sample collection periodically for pharmacological studies. Samples are analyzed for everolimus blood levels and correlated with 18FDG uptake suppression in tumor and normal brain via LC-MSMS. Previously collected tumor tissue are analyzed for protein biomarkers including PTEN gene expression levels via fluorescence in situ hybridization (FISH) and immunohistochemistry (IHC) and phosphorylation on Ser473 and Ser308 of Akt and MGMT expression and promoter methylation via IHC. Samples are also analyzed for DNA sequencing. Some samples are banked for future studies.

After completion of study treatment, patients are followed every 2 months for 1 year, every 3 months for 1 year, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 138 patients (24 patients in phase I and 114 patients in phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Glioblastoma multiforme (grade 4 astrocytoma)
  * Other grade 4 astrocytoma variants (e.g., giant cell)

    * No grade 4 oligodendrogliomas or oligoastrocytomas
  * Gliosarcoma
* Newly diagnosed disease
* Measurable disease ≥ 1 cm³ (phase I patients only)
* Some patients may be registered on protocol NCCTG-947252
* No oligodendrogliomas or oligoastrocytomas

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* ANC ≥ 1,500/μL
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/μL
* Total bilirubin ≤ 2.5 x institutional upper limit of normal (ULN)
* Serum total cholesterol < 350 mg/dL
* Serum total triglycerides < 400 mg/dL
* AST ≤ 2.5 x ULN
* Creatinine ≤ 1.5 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 60 days after completion of study therapy
* Must be willing to undergo 2 mandatory research PET or PET/CT scans (all MCR and MCJ patients in phase I and MCR only patients in phase II)
* Must be willing to abstain from eating or drinking grapefruit or grapefruit juice during study treatment
* Must be willing to follow a diet low in fat and cholesterol while taking everolimus
* Must be willing to have imaging scans submitted for central review
* Ability to understand and willingness to sign a written informed consent

Exclusion criteria:

* Other active cancers requiring therapy to control disease or prior cancer diagnoses which pose a greater than 30% risk of death within the next 2 years
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active uncontrolled peptic ulcer disease
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing, uncontrolled, or active (acute or chronic) infection or disorder
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Severely impaired lung function
  * Uncontrolled diabetes (fasting serum glucose > 2 x ULN) OR diabetes that would interfere with the performance of the FDG-PET/CT or FDG-PET scans
  * Liver disease (e.g., cirrhosis, chronic active hepatitis, chronic persistent hepatitis, or history of hepatitis B)
* Known HIV positivity
* Positive hepatitis B antigen (HBsAg) or hepatitis C serology (HCV) tests
* Any history of allergy or intolerance to dacarbazine (DTIC)
* Significant traumatic injury within the past 21 days
* Severe allergy to sulfa medications
* Inability to tolerate levofloxacin with dapsone or pentamidine (inhaled or IV)

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* At least 1 week, but no more than 6 weeks since prior surgical resection or biopsy
* Must comply with antibiotic prophylaxis with either trimethoprim/sulfamethoxazole (daily or 3 times per week), oral dapsone (daily) combined with daily levofloxacin, or monthly pentamidine (inhaled or IV) combined with daily levofloxacin

Exclusion criteria:

* Prior chemotherapy for any brain tumor
* Prior temozolomide or mTOR inhibitor therapies
* Any prior cranial radiotherapy
* Planned immunization with attenuated live vaccines ≤ 7 days prior to and during study period
* At least 21 days since prior major surgery (excluding neurosurgical biopsy, resection of brain tumor, or treatment of immediate post-neurosurgical complication [e.g., intracranial hematoma])
* Concurrent or prior treatment for this cancer with any other investigational agents
* Concurrent enzyme-inducing anticonvulsants (EIACs) or other strong inducers of CYP3A4 (i.e., carbamazepine, phenytoin, phenobarbital/primidone, rifabutin, rifampin, or St. John's wort)
* Concurrent therapeutic doses of warfarin

  * Low molecular weight heparin is allowed
* Concurrent systematic leukocyte growth factors (e.g., G-CSF or GM-CSF), except for the treatment of severe neutropenia
* Concurrent drugs or substances known to inhibit or induce CYP3A
* Other concurrent chronic treatment with immunosuppressive agents except dexamethasone
* Other concurrent anticancer agents
* Concurrent live vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jann N. Sarkaria, MD, Study Chair — Mayo Clinic
Locations (178):
- United States (178):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Mercy Clinic Cancer and Hematology - Rolla, Rolla, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Ma D, Galanis E, Schiff D, et al.: NCCTG N057K phase II trial of everolimus, temozolomide, and radiotherapy in patients with newly diagnosed glioblastoma: A North Central Cancer Treatment Group trial. [Abstract] J Clin Oncol 30 (Suppl 15): A-2031, 2012.
- [Result] Sarkaria JN, Galanis E, Wu W, Peller PJ, Giannini C, Brown PD, Uhm JH, McGraw S, Jaeckle KA, Buckner JC. North Central Cancer Treatment Group Phase I trial N057K of everolimus (RAD001) and temozolomide in combination with radiation therapy in patients with newly diagnosed glioblastoma multiforme. Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):468-75. doi: 10.1016/j.ijrobp.2010.05.064. Epub 2010 Sep 23. PMID 20864273
- [Result] Sarkaria JN, Peller PJ, Galanis E, et al.: FLT-PET analysis of early response to everolimus in newly diagnosed glioblastoma patients enrolled on NCCTG N057K. [Abstract] J Clin Oncol 29 (Suppl 15): A-e12501, 2011.

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Cohort/Dose Level 1 (30 mg RAD001): Cycle 1: Everolimus 30 mg days 1, 8, and weekly through radiation therapy (RT). Starting between day 8 and 15 RT was 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Everolimus. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Everolimus 30 mg/week (Days 1, 8, 15 and 22 for each cycle, until progression). Prophylaxis for pneumocystis carinii pneumonia (PCP) was required starting cycle 1 day1.
- Phase I: Cohort/Dose Level 2 (50 mg RAD001): Cycle 1: Everolimus 50 mg days 1, 8, and weekly through radiation therapy (RT). Starting between day 8 and 15 RT was 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Everolimus. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Everolimus 50 mg/week (Days 1, 8, 15 and 22 for each cycle, until progression). Prophylaxis for pneumocystis carinii pneumonia (PCP) was required starting cycle 1 day1.
- Phase 1: Cohort/Dose Level 3 (70 mg RAD001); Phase II: Cycle 1: Everolimus 70 mg days 1, 8, and weekly through radiation therapy (RT). Starting between day 8 and 15 RT was 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Everolimus. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Everolimus 70 mg/week (Days 1, 8, 15 and 22 for each cycle, until progression). Prophylaxis for pneumocystis carinii pneumonia (PCP) was required starting cycle 1 day1.
Period: Overall Study
Arm/Group | Phase I: Cohort/Dose Level 1 (30 mg RAD001) | Phase I: Cohort/Dose Level 2 (50 mg RAD001) | Phase 1: Cohort/Dose Level 3 (70 mg RAD001) | Phase II
Started | 6 | 6 | 6 | 104
Completed | 6 | 6 | 6 | 100
Not Completed | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Ineligible | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Cycle 1: Everolimus (either: 30, 50, or 70 mg) days 1, 8, and weekly through radiation therapy (RT). Starting between day 8 and 15 RT was 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Everolimus. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Everolimus (either: 30, 50, or 70 mg)/week (Days 1, 8, 15 and 22 for each cycle, until progression). Prophylaxis for pneumocystis carinii pneumonia (PCP) was required starting cycle 1 day1.
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 18 | 104 | 122
Age, Continuous [Median (Full Range); unit: years] | 57.5 [23 to 74] | 61 [23 to 81] | 60.5 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 50 | 59
  Male | 9 | 54 | 63
Region of Enrollment [Number; unit: participants]
  United States | 18 | 104 | 122

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Everolimus (RAD001) in Combination With Temozolomide (TMZ) and 3D-conformal Radiotherapy (RT) or Intensity-modulated Radiotherapy (IMRT) Followed by Adjuvant TMZ With or Without RAD001 (Phase I)
Description: Patients were assessed during RT for dose-limiting toxicities (DLT), which were defined as failure to deliver greater than 75% of the planned doses of TMZ or RAD001 during RT, interruption of RT for more than 5 days because of toxicity, or the following: >= Grade 3 diarrhea or skin rash; >= Grade 4 neutropenia, leukopenia, or thrombocytopenia; >= Grade 4 hypertriglyceridemia, hypercholesterolemia, or hyperglycemia despite optimal medial management, other >= 3 non-hematologic events; or >= Grade 4 radiation dermatitis. Maximum tolerated dose (MTD) was defined a priori as the highest dose level at which 0 or 1 of 6 patients developed DLTs. The number of patients who developed DLTs are reported here by dose level, with the MTD reported in the statistical analysis section.
Time Frame: Up to 49 days
Population: Eighteen patients were enrolled in Phase I of the study to determine the maximum tolerated dose (MTD). The dosage of RAD001 was escalated in cohorts of 6 patients.
Measure: Number; unit: participants who developed DLTs
Groups:
- Phase I: Dose Level 0: Cycle 1: Everolimus 30 mg days 1, 8, and weekly through radiation therapy (RT). Starting between day 8 and 15 RT was 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Everolimus. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Everolimus 30 mg/week (Days 1, 8, 15 and 22 for each cycle, until progression). Prophylaxis for pneumocystis carinii pneumonia (PCP) was required starting cycle 1 day1.
- Phase I: Dose Level 1: Cycle 1: Everolimus 50 mg days 1, 8, and weekly through radiation therapy (RT). Starting between day 8 and 15 RT was 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Everolimus. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Everolimus 50 mg)/week (Days 1, 8, 15 and 22 for each cycle, until progression). Prophylaxis for pneumocystis carinii pneumonia (PCP) was required starting cycle 1 day1.
- Phase I: Dose Level 2: Cycle 1: Everolimus 70 mg days 1, 8, and weekly through radiation therapy (RT). Starting between day 8 and 15 RT was 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Everolimus. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Everolimus 70 mg/week (Days 1, 8, 15 and 22 for each cycle, until progression). Prophylaxis for pneumocystis carinii pneumonia (PCP) was required starting cycle 1 day1.
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2
Number analyzed (Participants) | 6 | 6 | 6
participants who developed DLTs | 1 | 1 | 1
Statistical Analysis 1: Comparison: Phase I: Dose Level 0 vs Phase I: Dose Level 1 vs Phase I: Dose Level 2; Test type: Superiority or Other; Maximum Tolerated Dose (mg) = 70

2. Primary Outcome: Overall Survival at 12 Months (Phase II)
Description: The primary endpoint is overall survival at 12 months (OS12) after entry into this study. The proportion of successes will be estimated using the binomial point estimator (number of successes divided by the total number of evaluable patients) and the binomial 95% confidence interval estimated. A patient who is evaluable and survive more than 12 months (i.e. 365 days or more) after start of therapy will be classified as a "success". Patients who die within 12 months after start of therapy will be considered to have "failed".
Time Frame: at 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase II
Number analyzed (Participants) | 100
proportion of participants | 0.64 [0.553 to 0.741]

3. Secondary Outcome: Response Rate, as Measured in Patients Receiving FLT-PET Imaging (Phase II)
Description: The response rate is defined as the percentage of patients receiving F-fluorothymidine positron emission tomography (FLT-PET) imaging whose cancer shrinks or disappears after treatment. A reduction in standardized uptake value (SUV) of 30% or greater in the T1-post-gadolinium scan volume of interest (T1-gad VOI) or the total tumor VOI will be considered a responsive tumor.
Time Frame: Up to 5 years
Population: Of the 11 patients with measurable residual disease and pre-everolimus FLT-PET imaging, 2 did not have a second FLT-PET scan performed due to technical difficulties with FLT production, leaving 9 patients who could be assessed for changes in FLT uptake.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 9
percentage of participants | 44.4 [15.3 to 77.3]

4. Secondary Outcome: Time to Progression (Phase II)
Description: Time-to-disease progression is defined as the time from start of study therapy to documentation of disease progression. Patients who die without documentation of progression will be considered to have had tumor progression at the time of death unless there is documented evidence that no progression occurred before death. Patients who fail to return for evaluation after beginning therapy will be censored for progression on the last day of therapy. Patients who experience major treatment violations will be censored for progression on the date of treatment violation occurred. The time-to-progression distribution will be estimated using the Kaplan-Meier method. Progression is defined as at least a 25% increase in product of perpendicular diameters of contrast enhancement or mass or unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians or appearance of new lesions.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 100
months | 6.4 [5.4 to 9.0]

5. Secondary Outcome: Progression-free-survival at 6 Months (Phase II)
Description: Progression-free-survival at 6 months: is the proportion of patients alive and progression-free at 6 months after start of regimen. This proportion will be estimated using the binomial point estimator and the binomial 95% confidence interval estimated. Progression is defined as at least a 25% increase in product of perpendicular diameters of contrast enhancement or mass or unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians or appearance of new lesions.
Time Frame: at 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase II
Number analyzed (Participants) | 100
proportion of participants | 0.52 [0.431 to 0.628]

6. Secondary Outcome: Overall Survival Time
Description: Overall survival: The overall survival or survival time is defined as the time from registration to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier method.
Time Frame: Up to 15 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 100
months | 15.8 [13.0 to 20.3]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed weekly during Cycle 1, at the end of RT, prior to cycles 3-8, and during treatment with everolimus only until progression (Cycles ≥9). Only patients who had completed one cycle of treatment and completed an adverse event form were included in this adverse event table; Up to 5 years.
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized until September 30, 2010. CTCAE version 4.0 will be utilized for expedited adverse event reporting only, beginning October 1, 2010. All appropriate treatment areas should have access to a copy of the CTCAE v4.0.
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 5/18 | 32/101
Other Adverse Events (participants affected / at risk) | 18/18 | 99/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=18) | Phase II (N=101)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (2) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (2) | 3 (4)
Fever (General disorders) | 0 (0) | 2 (2)
Localized edema (General disorders) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Bilirubin increased (Investigations) | 1 (2) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (2) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (2) | 10 (11)
Platelet count decreased (Investigations) | 1 (2) | 9 (9)
Serum cholesterol increased (Investigations) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=18) | Phase II (N=101)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 9 (17)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 3 (3)
Watering eyes (Eye disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 7 (11) | 35 (79)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 6 (6)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (20) | 68 (166)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Edema limbs (General disorders) | 0 (0) | 7 (11)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (6) | 45 (83)
Fever (General disorders) | 0 (0) | 2 (2)
Irritability (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (4) | 3 (3)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 3 (3)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (3)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 6 (11)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (8)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 5 (9) | 16 (30)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (19) | 42 (108)
Platelet count decreased (Investigations) | 15 (40) | 64 (187)
Serum cholesterol increased (Investigations) | 16 (80) | 80 (359)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 5 (21)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 14 (17)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 12 (15)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Serum triglycerides increased (Metabolism and nutrition disorders) | 13 (57) | 70 (286)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 1 (2)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 14 (19)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (4)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 4 (4)
Speech disorder (Nervous system disorders) | 1 (1) | 6 (20)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1) | 7 (11)
Tremor (Nervous system disorders) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (5)
Confusion (Psychiatric disorders) | 1 (1) | 6 (8)
Depression (Psychiatric disorders) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 6 (6)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 38 (97)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 29 (63)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (11) | 48 (105)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Thrombosis (Vascular disorders) | 2 (2) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes